CLINICAL TRIAL: NCT00623454
Title: A Randomized Controlled Trial of Cognitive Behavioural Therapy for Non-cardiac Chest Pain and Palpitations.
Brief Title: Non Cardiac Chest Pain and Benign Palpitations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4.2006.1110 (REK)
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Anxiety/Depression in Cardiological Unit
Keywords: anxiety; panic disorder; chest pain; palpitations
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Chest Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive behaviour therapy — Three hours with cognitive therapy focusing on the chest pain and palpitations.

SUMMARY:
All Patients between 18 and 65 years are asked 6 month after investigation for chest pain or palpitation at Cardiological Out-patient Clinic, Molde Hospital, about if they still have symptoms of chest pain or palpitation. If they still have some of the symptoms they are invited to participate in a coping course to learn a better way to deal with their symptoms.

The coping course consist of three sessions of cognitive behaviour therapy.

ELIGIBILITY:
Inclusion Criteria:

* investigated for chest pain or palpitation 6 month ago at Cardiological Out-patient Clinic, Molde Hospital
* suffer of chest pain or palpitations

Exclusion Criteria:

* do not speak norwegian properly
* mentally retarded
* psychosis last 6 month
* current alcohol or drug misuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Body sensation questionnaire (BSQ) | end of treatment, after 3 month and after 12 month
Beck Depression Inventory (BDI) | end of treatment, after 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Egil Jonsbu, MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Cardiological Out-patient Clinic, Molde, Molde, Norway

REFERENCES:
- [Result] Jonsbu E, Dammen T, Morken G, Martinsen EW. Patients with noncardiac chest pain and benign palpitations referred for cardiac outpatient investigation: a 6-month follow-up. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):406-12. doi: 10.1016/j.genhosppsych.2010.03.003. Epub 2010 Apr 13. PMID 20633745